CLINICAL TRIAL: NCT02969655
Title: A 52-week, Phase III, Double-blind, Active-controlled, Parallel-group, Multi-center Study to Evaluate Efficacy and Safety of Daprodustat Compared to Darbepoetin Alfa in Japanese Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease Who Are Currently ESA Users
Brief Title: A Study to Evaluate Efficacy and Safety of Daprodustat Compared to Darbepoetin Alfa in Japanese Hemodialysis (HD)-Dependent Subjects With Anemia Associated With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201754
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Anaemia
Keywords: Safety; Efficacy; Daprodustat; Chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daprodustat (Experimental): Subjects will receive oral daprodustat once daily and intravenous (IV) darbepoetin alfa placebo once weekly for 52 weeks
  Interventions: Drug: Daprodustat small; Drug: Daprodustat large; Drug: Darbepoetin alfa placebo
- Darbepoetin alfa (Active Comparator): Subjects will receive IV darbepoetin alfa once weekly and oral daprodustat placebo once daily for 52 weeks
  Interventions: Drug: Daprodustat small placebo; Drug: Daprodustat large placebo; Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Daprodustat small — Available as 7.0 millimeter (mm) round, standard biconvex, white film coated tablets containing 1 mg, 2 mg, or 4 mg of daprodustat as active ingredient
  Arms: Daprodustat
Drug: Daprodustat small placebo — Available as 7.0 mm round, standard biconvex, white film coated tablets containing no daprodustat
  Arms: Darbepoetin alfa
Drug: Daprodustat large — Available as 9.0 mm round, standard biconvex, white film coated tablets containing 6 mg of daprodustat as active ingredient
  Arms: Daprodustat
Drug: Daprodustat large placebo — Available as 9.0 mm round, standard biconvex, white film coated tablets containing no daprodustat
  Arms: Darbepoetin alfa
Drug: Darbepoetin alfa — Available as 0.5 mL plastic prefilled syringes (PFS) for IV injection each containing 10, 15, 20, 30, 40 or 60 mcg of darbepoetin alfa in a clear and colorless solution.
  Arms: Darbepoetin alfa
Drug: Darbepoetin alfa placebo — Available as 0.5 mL plastic PFS for IV injection containing no darbepoetin alfa in a clear and colorless solution.
  Arms: Daprodustat

SUMMARY:
Daprodustat is a drug that is currently being developed as a treatment for renal anemia . This study is to evaluate the efficacy and safety of daprodustat following a switch from erythropoiesis-stimulating agent (ESA) in Japanese HD subjects with renal anemia who are currently treated with ESA. The primary objective is to demonstrate non-inferiority of daprodustat to darbepoetin alfa. This study is a 52-week, Phase III, double-blind, active-controlled, parallel-group, multi-center study. The total duration of the study will be approximately 58 weeks including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria

* Age (informed consent): >=20 years of age
* Dialysis: On HD or hemodiafiltration (HDF) given three times weekly for at least 12 weeks prior to screening
* ESAs: Use of one and the same ESA for 10 weeks prior to screening
* ESA dose: Darbepoetin alfa 10 to 60 μg per week, epoetin (including biosimilars) <=9000 international units (IU) per week, or epoetin beta pegol <=250 μg per 4 weeks
* Hgb:>=9.5 g/dL and <=12.5 g/dL. Determined at the site using an Hgb analyzer
* Iron parameters: Ferritin >100 nanogram (ng)/millilitre (mL) or transferrin saturation (TSAT) >20 percent (screening verification only)
* Gender (screening verification only): Female or male

Females: Not pregnant [demonstrated to be negative for human chorionic gonadotropin (hCG) in serum], not breast-feeding, and meet at least one of the following:

• Females of non-childbearing potential are defined as follows:

Pre-menopausal with at least one of the following and no plans to utilise assisted reproductive techniques (e.g., in vitro fertilisation or donor embryo transfer):

* History of bilateral tubal ligation or salpingectomy
* History of hysteroscopic tubal occlusion and postoperatively documented bilateral tubal obstruction
* History of hysterectomy
* History of bilateral oophorectomy Postmenopausal defined as A) females 60 years of age or older or B) In females < 60 years of age, 12 months of spontaneous amenorrhea [in questionable cases a blood sample with postmenopausal follicle stimulating hormone (FSH) and estradiol concentrations is confirmatory (see separately specified reference ranges)]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the most effective contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

  • Females of childbearing potential must agree to comply with one of the contraception methods listed as requirements in "GlaxoSmithKline (GSK) Listing of Most Effective Contraceptive Methods for Females of Childbearing Potential from 28 days prior to the first dose of study medication until the completion of the follow-up visit.
* Informed consent: Written informed consent, including adherence to the requirements and conditions specified in the consent form and the protocol, must be obtained from each subject.

Exclusion Criteria

CKD-related criteria

* Kidney transplant: Planned living-related kidney transplant during the study

Anemia-related criteria

* Aplasia: History of bone-marrow hypoplasia or pure red cell aplasia
* Other causes of anemia: pernicious anemia, thalassemia, sickle cell anemia, or myelodysplastic syndromes
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within 10 weeks prior to screening or during a period from screening to Day 1

Cardiovascular disease-related criteria

* Myocardial infarction, acute coronary syndrome, stroke, or transient ischemic attack: Diagnosed within 10 weeks prior to screening or during a period from screening to Day 1
* Heart failure: Chronic Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system
* Corrected QT (QTc) Interval (screening verification only): QTc >500 milliseconds (msec); or QTc >530 msec in subjects with bundle branch block Note: QT interval corrected using the Bazett's formula (QTcB) will be used, and electrocardiogram (ECG) can be mechanically or manually read

Other disease-related criteria:

* Liver disease (if any of the following occurs):

  * Alanine transaminase (ALT) >2 upper limit of normal (ULN)
  * Bilirubin >1.5×ULN (isolated bilirubin >1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35 percent)
  * Current unstable active liver or biliary disease (generally defined by the onset of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, persistent jaundice, or cirrhosis)
* Malignancy: History of malignancy within 2 years prior to screening, currently receiving treatment for cancer, or complex kidney cyst >3 centimeters (cm) (II F, III or IV based on the Bosniak classification)

Concomitant medication and other study treatment-related criteria

* Iron: Planned use of intravenous iron during the screening phase or during a period from Day 1 to Week 4
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
* Drugs and supplements: Use or planned use of any prescription or non-prescription drugs or dietary supplements that are prohibited during the study period [prohibited medications: strong inducers and inhibitor of Cytochrome P450 (CYP) 2C8].
* Prior investigational product exposure: Use of an investigational agent within 30 days or five half lives of the investigational agent (whichever is longer)
* Prior treatment with daprodustat: Any prior treatment with daprodustat for a treatment duration of >30 days

General health-related criteria

* Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator (or subinvestigator) considers would put the subject at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Japan (22):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20737

REFERENCES:
- [Background] Akizawa T, Nangaku M, Yonekawa T, Okuda N, Kawamatsu S, Onoue T, Endo Y, Hara K, Cobitz AR. Efficacy and Safety of Daprodustat Compared with Darbepoetin Alfa in Japanese Hemodialysis Patients with Anemia: A Randomized, Double-Blind, Phase 3 Trial. Clin J Am Soc Nephrol. 2020 Aug 7;15(8):1155-1165. doi: 10.2215/CJN.16011219. Epub 2020 Jul 28. PMID 32723804
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 centers, contracted in Japan, enrolled and randomized participants. A total of 271 participants were enrolled and randomized in this study.
Pre-assignment Details: A total of 332 participants were screened of which 61 failed screening reasons being participants did not meet inclusion/exclusion criteria (48), physician decision (3) and withdrawn by participant (10), hence 271 participants were enrolled and randomized.
Groups:
- Daprodustat: Participants received oral daprodustat tablets (1, 2, 4, 6, 8, 12, 18 and 24 milligrams [mg] as recommended) once daily and intravenous (IV) darbepoetin alfa placebo injection (0.5 milliliter prefilled syringes containing no darbepoetin alfa) once weekly for 52 weeks.
- Darbepoetin Alfa: Participant received IV darbepoetin alfa injection (10,15,20,30,40 and 60 micrograms [ug] as recommended) once weekly and oral daprodustat placebo tablets (small and large tablets containing no daprodustat) once daily for 52 weeks.
Period: Overall Study
Arm/Group | Daprodustat | Darbepoetin Alfa
Started | 136 | 135
Completed | 115 | 120
Not Completed | 21 | 15
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 4 | 3
Not completed — Protocol-specified withdrawal criteria | 4 | 2
Not completed — Adverse Event | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 136 | 135 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (10.30) | 63.5 (10.54) | 63.8 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 91 | 89 | 180
Race/Ethnicity, Customized [Number; unit: Count of participants]
  Asian - Japanese heritage | 136 | 135 | 271

OUTCOME MEASURES:

1. Primary Outcome: Mean Hemoglobin (Hgb) During the Primary Efficacy Evaluation Period (Weeks 40 to 52)
Description: The mean hemoglobin during the Evaluation Period was estimated by a statistical model.
Time Frame: Weeks 40 to 52
Population: Intent to treat (ITT) Population comprised of all randomized participants who had a Baseline and at least one post Baseline schedule Hgb assessment.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Grams per deciliter (g/dL) | 10.89 (0.062) | 10.83 (0.060)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was established if the lower limit of the 95% CI was greater than -1.0 g/dL. Even if the 95% CI for the difference was completely negative (i.e. lied fully within the range -1.0 to <0 g/dL) non-inferiority was concluded on condition that the mean Hgb estimated in the daprodustat group was within the target range; p < .0001, Mixed model repeated measures (MMRM) — The p value on this table is one-sided and calculated for the non-inferiority assessment; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.11 to 0.23] — Analysis was performed by a MMRM with covariates of treatment, Baseline Hgb, visit, treatment-by-visit interaction, Baseline-by-visit interaction

2. Secondary Outcome: Percentage of Participants With Mean Hgb in the Target Range (10.0-12.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52)
Description: The percentage of participants with observed mean Hgb within the target range during the primary efficacy evaluation period was summarized. Odds ratio was estimated using a logistic regression and provided along with its 95% CI and a one-sided p-value.
Time Frame: Weeks 40 to 52
Population: Modified Intent to treat (mITT) comprised of all ITT participants who had at least one Hgb measurement during the evaluation period.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 120 | 125
Percentage of participants
  Responder | 88 | 90
  Non-responder | 13 | 10
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7442, Regression, Logistic — The p value on this table is one-sided and calculated for the superiority assessment; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.34 to 1.71] — Analysis was performed by logistic regression with covariates of treatment and Baseline Hgb

3. Secondary Outcome: Change From Baseline in Hgb (Hgb Increase Rate) at Week 4
Description: Change from Baseline was calculated as the post-dose Week 4 visit value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
g/dL | -0.42 (0.898) | 0.08 (0.525)

4. Secondary Outcome: Percentage of Participants by Hgb Change From Baseline Category at Week 4
Description: Percentage of participants within each category were provided only for daprodustat and the categories were classified into 6 (i.e., <=-2, >-2 to -1, >-1 to 0, >0 to 1, >1 to 2, >2 grams per deciliter [g/dL]). In addition, 'within 1.0 g/dL (i.e., <=-1 and >=1) and over 2.0 g/dL (i.e., <-2 and >2) categories were provided.
Time Frame: Week 4
Population: ITT Population. Data for Darbepoetin alfa group could not be collected as comparison was not reasonable because of the difference in dose adjustment frequency.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat
Number analyzed (Participants) | 133
Percentage of participants
  <= -2.0 | 5
  > -2.0 and <= -1.0 | 21
  > -1.0 and <= 0 | 44
  > 0 and <= 1.0 | 27
  > 1.0 and <= 2.0 | 4
  > 2.0 | 0
  within +/- 1.0 | 75
  over +/- 2.0 | 5

5. Secondary Outcome: Distribution of Daprodustat Dose Level by Visit
Description: Distribution of dose level by visit for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented for Daprodustat. Median along with the interquartile range (25th and 75th percentile) has been presented.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44, and 48)
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Median (Inter-Quartile Range); unit: milligrams per day (mg/day)
Arm/Group | Daprodustat
Number analyzed (Participants) | 133
milligrams per day (mg/day)
  Day 1, n=133 | 4.0 [4.0 to 4.0]
  Week 4, n=133 | 4.0 [4.0 to 6.0]
  Week 8, n=126: number analyzed (Participants) | 126
  Week 8, n=126 | 4.0 [4.0 to 6.0]
  Week 12, n=125: number analyzed (Participants) | 125
  Week 12, n=125 | 6.0 [4.0 to 6.0]
  Week 16, n=123: number analyzed (Participants) | 123
  Week 16, n=123 | 6.0 [4.0 to 8.0]
  Week 20, n=123: number analyzed (Participants) | 123
  Week 20, n=123 | 6.0 [4.0 to 8.0]
  Week 24, n=123: number analyzed (Participants) | 123
  Week 24, n=123 | 6.0 [4.0 to 8.0]
  Week 28, n=123: number analyzed (Participants) | 123
  Week 28, n=123 | 6.0 [4.0 to 8.0]
  Week 32, n=122: number analyzed (Participants) | 122
  Week 32, n=122 | 6.0 [4.0 to 8.0]
  Week 36, n=121: number analyzed (Participants) | 121
  Week 36, n=121 | 6.0 [4.0 to 8.0]
  Week 40, n=119: number analyzed (Participants) | 119
  Week 40, n=119 | 6.0 [4.0 to 8.0]
  Week 44, n=117: number analyzed (Participants) | 117
  Week 44, n=117 | 6.0 [4.0 to 8.0]
  Week 48, n=117: number analyzed (Participants) | 117
  Week 48, n=117 | 6.0 [4.0 to 8.0]

6. Secondary Outcome: Distribution of Darbepoetin Alfa Dose Level by Visit
Description: Distribution of dose level by visit for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented for Darbepoetin Alfa. Median along with the interquartile range (25th and 75th percentile) has been presented.
Time Frame: Day 1, Weeks 2,4,6,8,10,12,14,16,18,20,22,24,26,28,30,32,34,36,38,40,42,44,46,48, and 50
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: micrograms per week (ug/week)
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 134
micrograms per week (ug/week)
  Day 1, n=134 | 15.0 [15.0 to 30.0]
  Week 2. n=134 | 15.0 [15.0 to 30.0]
  Week 4, n=134 | 15.0 [10.0 to 30.0]
  Week 6, n=133: number analyzed (Participants) | 133
  Week 6, n=133 | 15.0 [10.0 to 30.0]
  Week 8, n=131: number analyzed (Participants) | 131
  Week 8, n=131 | 15.0 [10.0 to 30.0]
  Week 10, n=129: number analyzed (Participants) | 129
  Week 10, n=129 | 15.0 [10.0 to 30.0]
  Week 12, n=129: number analyzed (Participants) | 129
  Week 12, n=129 | 15.0 [10.0 to 30.0]
  Week 14, n=129: number analyzed (Participants) | 129
  Week 14, n=129 | 15.0 [10.0 to 30.0]
  Week 16, n=129: number analyzed (Participants) | 129
  Week 16, n=129 | 15.0 [10.0 to 30.0]
  Week 18, n=129: number analyzed (Participants) | 129
  Week 18, n=129 | 15.0 [10.0 to 30.0]
  Week 20, n=129: number analyzed (Participants) | 129
  Week 20, n=129 | 15.0 [10.0 to 30.0]
  Week 22, n=128: number analyzed (Participants) | 128
  Week 22, n=128 | 15.0 [10.0 to 30.0]
  Week 24, n=129: number analyzed (Participants) | 129
  Week 24, n=129 | 15.0 [10.0 to 30.0]
  Week 26, n=129: number analyzed (Participants) | 129
  Week 26, n=129 | 15.0 [10.0 to 30.0]
  Week 28, n=127: number analyzed (Participants) | 127
  Week 28, n=127 | 15.0 [10.0 to 30.0]
  Week 30, n=128: number analyzed (Participants) | 128
  Week 30, n=128 | 15.0 [10.0 to 30.0]
  Week 32, n=127: number analyzed (Participants) | 127
  Week 32, n=127 | 15.0 [10.0 to 30.0]
  Week 34, n=127: number analyzed (Participants) | 127
  Week 34, n=127 | 15.0 [10.0 to 30.0]
  Week 36, n=127: number analyzed (Participants) | 127
  Week 36, n=127 | 15.0 [10.0 to 30.0]
  Week 38, n=127: number analyzed (Participants) | 127
  Week 38, n=127 | 15.0 [10.0 to 30.0]
  Week 40, n=125: number analyzed (Participants) | 125
  Week 40, n=125 | 15.0 [10.0 to 30.0]
  Week 42, n=125: number analyzed (Participants) | 125
  Week 42, n=125 | 15.0 [10.0 to 30.0]
  Week 44, n=125: number analyzed (Participants) | 125
  Week 44, n=125 | 15.0 [10.0 to 30.0]
  Week 46, n=125: number analyzed (Participants) | 125
  Week 46, n=125 | 15.0 [10.0 to 30.0]
  Week 48, n=124: number analyzed (Participants) | 124
  Week 48, n=124 | 15.0 [10.0 to 30.0]
  Week 50, n=122: number analyzed (Participants) | 122
  Week 50, n=122 | 15.0 [10.0 to 30.0]

7. Secondary Outcome: Duration of Treatment Interruption Due to Hgb >13 g/dL
Description: Duration of treatment interruption due to Hgb >13 g/dL for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented for the daprodustat group.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the time of assessment were used for analysis. Summary data for Darbepoetin alfa group could not be collected as comparison was not reasonable because of the difference in dose adjustment frequency. Median along with inter quartile range (25th and 75th percentile) have been presented.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Daprodustat
Number analyzed (Participants) | 3
Days | 28.0 [28.0 to 56.0]

8. Secondary Outcome: Number of Dose Adjustments for Daprodustat
Description: Number of dose adjustments has been presented only for daprodustat.
Time Frame: Up to Week 52
Population: ITT Population. Summary data for Darbepoetin alfa group could not be collected as comparison was not reasonable because of the difference in dose adjustment frequency.
Measure: Median (Full Range); unit: Dose adjustments
Arm/Group | Daprodustat
Number analyzed (Participants) | 133
Dose adjustments | 2.0 [0 to 6]

9. Secondary Outcome: Hgb Values at Each Assessment Visit
Description: Hgb values at each assessment visit for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented.
Time Frame: Baseline (Day 1), Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
g/dL
  Baseline (Day 1), n=133, 134 | 10.94 (0.770) | 10.82 (0.732)
  Week 4, n=133, 134 | 10.52 (0.984) | 10.90 (0.829)
  Week 8, n=127, 132: number analyzed (Participants) | 127 | 132
  Week 8, n=127, 132 | 10.50 (1.069) | 11.01 (0.824)
  Week 12, n=125, 129: number analyzed (Participants) | 125 | 129
  Week 12, n=125, 129 | 10.53 (0.989) | 11.09 (0.753)
  Week 16, n=124, 129: number analyzed (Participants) | 124 | 129
  Week 16, n=124, 129 | 10.57 (0.970) | 10.92 (0.862)
  Week 20, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 20, n=123, 129 | 10.85 (0.784) | 10.95 (0.830)
  Week 24, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 24, n=123, 129 | 11.01 (0.718) | 10.92 (0.859)
  Week 28, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 28, n=123, 129 | 10.97 (0.748) | 10.86 (0.872)
  Week 32, n=122, 127: number analyzed (Participants) | 122 | 127
  Week 32, n=122, 127 | 11.10 (0.829) | 10.96 (0.820)
  Week 36, n=121, 127: number analyzed (Participants) | 121 | 127
  Week 36, n=121, 127 | 11.12 (0.827) | 10.91 (0.847)
  Week 40, n=120, 125: number analyzed (Participants) | 120 | 125
  Week 40, n=120, 125 | 10.97 (0.860) | 10.90 (0.835)
  Week 44, n=117, 125: number analyzed (Participants) | 117 | 125
  Week 44, n=117, 125 | 10.98 (0.912) | 10.87 (0.904)
  Week 48, n=117, 124: number analyzed (Participants) | 117 | 124
  Week 48, n=117, 124 | 10.94 (0.893) | 10.76 (0.830)
  Week 52,n=115, 120: number analyzed (Participants) | 115 | 120
  Week 52,n=115, 120 | 10.79 (0.807) | 10.79 (0.841)

10. Secondary Outcome: Change From Baseline in Hgb Values at Each Assessment Visit
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calcuated as the post-dose visit value minus the Baseline value. Change from Baseline Hgb values at each assessment visit for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented.
Time Frame: Baseline (Day 1) and Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
g/dL
  Week 4, n=133, 134 | -0.42 (0.898) | 0.08 (0.525)
  Week 8, n=127, 132: number analyzed (Participants) | 127 | 132
  Week 8, n=127, 132 | -0.45 (1.178) | 0.20 (0.821)
  Week 12, n=125, 129: number analyzed (Participants) | 125 | 129
  Week 12, n=125, 129 | -0.42 (1.258) | 0.27 (1.021)
  Week 16, n=124, 129: number analyzed (Participants) | 124 | 129
  Week 16, n=124, 129 | -0.38 (1.348) | 0.09 (1.146)
  Week 20, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 20, n=123, 129 | -0.09 (1.161) | 0.12 (1.120)
  Week 24, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 24, n=123, 129 | 0.07 (1.106) | 0.10 (1.068)
  Week 28, n=123, 129: number analyzed (Participants) | 123 | 129
  Week 28, n=123, 129 | 0.03 (1.084) | 0.04 (1.080)
  Week 32, n=122, 127: number analyzed (Participants) | 122 | 127
  Week 32, n=122, 127 | 0.16 (1.119) | 0.14 (1.071)
  Week 36, n=121, 127: number analyzed (Participants) | 121 | 127
  Week 36, n=121, 127 | 0.17 (1.020) | 0.09 (1.041)
  Week 40, n=120, 125: number analyzed (Participants) | 120 | 125
  Week 40, n=120, 125 | 0.03 (1.060) | 0.10 (1.034)
  Week 44, n=117, 125: number analyzed (Participants) | 117 | 125
  Week 44, n=117, 125 | 0.03 (1.118) | 0.07 (1.019)
  Week 48, n=117, 124: number analyzed (Participants) | 117 | 124
  Week 48, n=117, 124 | -0.01 (1.164) | -0.04 (0.978)
  Week 52,n=115, 120: number analyzed (Participants) | 115 | 120
  Week 52,n=115, 120 | -0.16 (1.169) | 0.01 (1.019)

11. Secondary Outcome: Percentage of Participants Who Had Hgb Level Within the Target Range (10.0-12.0 g/dL) at Each Assessment Visit
Description: Percentage of participants with Hgb within the target range was summarized at each assessment visit by treatment group have been presented.
Time Frame: Baseline (Day 1) and Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Percentage of participants
  Baseline (Day 1), n=133, 134 | 79 | 87
  Week 4, n=133,134 | 65 | 80
  Week 8, n=127,132: number analyzed (Participants) | 127 | 132
  Week 8, n=127,132 | 65 | 84
  Week 12, n=125,129: number analyzed (Participants) | 125 | 129
  Week 12, n=125,129 | 66 | 86
  Week 16, n=124,129: number analyzed (Participants) | 124 | 129
  Week 16, n=124,129 | 64 | 80
  Week 20, n=123,129: number analyzed (Participants) | 123 | 129
  Week 20, n=123,129 | 82 | 81
  Week 24, n=123,129: number analyzed (Participants) | 123 | 129
  Week 24, n=123,129 | 85 | 81
  Week 28, n=123,129: number analyzed (Participants) | 123 | 129
  Week 28, n=123,129 | 85 | 82
  Week 32, n=122, 127: number analyzed (Participants) | 122 | 127
  Week 32, n=122, 127 | 79 | 80
  Week 36, n=121,127: number analyzed (Participants) | 121 | 127
  Week 36, n=121,127 | 78 | 78
  Week 40, n=120,125: number analyzed (Participants) | 120 | 125
  Week 40, n=120,125 | 77 | 80
  Week 44, n=117,125: number analyzed (Participants) | 117 | 125
  Week 44, n=117,125 | 74 | 82
  Week 48, n=117,124: number analyzed (Participants) | 117 | 124
  Week 48, n=117,124 | 77 | 79
  Week 52, n=115,120: number analyzed (Participants) | 115 | 120
  Week 52, n=115,120 | 77 | 80

12. Secondary Outcome: Percentage of Time in Hgb Target Range (10.0 to 12.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52)
Description: Percentage of time in Hgb target range (10.0 to 12.0 g/dL) during the primary efficacy evaluation period (Weeks 40 to 52) for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users has been presented.
Time Frame: Weeks 40 to 52
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 118 | 125
Percentage of time | 76.81 (30.387) | 80.23 (28.038)

13. Secondary Outcome: Number of Participants Who Had an Hgb Level of Less Than 7.5 g/dL
Description: If an initial Hgb value was less than 7.5 g/dL, measurement was repeated at the same study visit (using the same sample) to calculate the average. If the average met the Hgb stopping criteria, study treatment was permanently discontinued. Number of participants who had an Hgb level of less than 7.5 g/dL has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Percentage of participants | 0 | 0

14. Secondary Outcome: Number of Participants Who Had an Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Number of participants who had an Hgb increase of more than 2 g/dL over any 4 weeks for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users have been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Participants | 1 | 2

15. Secondary Outcome: Number of Participants Who Had an Hgb Level of More Than 13.0 g/dL
Description: Number of participants who had an Hgb increase of more than 13 g/dL for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users have been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Percentage of participants | 7 | 8

16. Secondary Outcome: Number of Episodes With Hgb Level of More Than 13.0 g/dL
Description: Number of episodes with Hgb level of more than 13.0 g/dL for hemodialysis-dependent participants with anemia associated with chronic kidney disease who were currently ESA users have been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Episodes
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 134
Episodes | 9 | 12

17. Secondary Outcome: Area Under Plasma Concentration Curve From Time Zero to 4 Hours (AUC [0 - 4]) of Plasma Daprodustat
Description: Blood samples for Pharmacokinetic (PK) analysis of daprodustat were collected as the time points provided. PK parameters were calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (version 6.3 or higher). NA indicates geometric co-efficient of variation could not be calculated as a single participant was analyzed. Data has been provided as a consolidated values for at all time-points (0,1,2,3,and 4 hours post-dose) as provided for a single value at Weeks 12 and 24 respectively. PK population comprised of all daprodustat-treated participants from whom PK samples were collected and analyzed. Data was not calculated for darbepoetin alfa group as the primary interest of analysis was Daprodustat and not comparator drug (darbepoetin alfa). Data is combined from Week 12 and Week 24 data.
Time Frame: 0, 1, 2, 3, and 4 hours post-dose at Week 12 and Week 24
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 125
Hours*nanograms per milliliter
  1 mg, n=8: number analyzed (Participants) | 8
  1 mg, n=8 | 27.57 (147.6)
  2 mg, n=24: number analyzed (Participants) | 24
  2 mg, n=24 | 44.52 (139.2)
  4 mg, n=91: number analyzed (Participants) | 91
  4 mg, n=91 | 72.68 (242.2)
  6 mg, n=61: number analyzed (Participants) | 61
  6 mg, n=61 | 140.58 (238.9)
  8 mg, n=38: number analyzed (Participants) | 38
  8 mg, n=38 | 170.41 (136.1)
  12 mg, n=17: number analyzed (Participants) | 17
  12 mg, n=17 | 150.53 (176.4)
  18 mg, n=5: number analyzed (Participants) | 5
  18 mg, n=5 | 488.93 (89.2)

18. Secondary Outcome: Maximum Concentration (Cmax) of Plasma Daprodustat
Description: Blood samples for PK analysis of daprodustat were collected as the time points provided. PK parameters were calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (version 6.3 or higher). Data has been provided as a consolidated values for at all time-points (0,1,2,3,and 4 hours post-dose) as provided for a single value at Weeks 12 and 24 respectively. Data was not calculated for darbepoetin alfa group as the primary interest of analysis was Daprodustat and not comparator drug (darbepoetin alfa). Data is combined from Week 12 and Week 24 data.
Time Frame: 0, 1, 2, 3, and 4 hours post-dose at Week 12 and Week 24
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 125
Nanograms per milliliter
  1 mg, n=8: number analyzed (Participants) | 8
  1 mg, n=8 | 16.11 (105.7)
  2 mg, n=24: number analyzed (Participants) | 24
  2 mg, n=24 | 25.16 (122.7)
  4 mg, n=91: number analyzed (Participants) | 91
  4 mg, n=91 | 42.45 (237.9)
  6 mg, n=61: number analyzed (Participants) | 61
  6 mg, n=61 | 83.60 (269.7)
  8 mg, n=38: number analyzed (Participants) | 38
  8 mg, n=38 | 105.71 (110.9)
  12 mg, n=17: number analyzed (Participants) | 17
  12 mg, n=17 | 108.58 (117.8)
  18 mg, n=5: number analyzed (Participants) | 5
  18 mg, n=5 | 306.61 (61.0)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from the start of study treatment until the follow-up contact (Day 1 up to Follow-up Visit [Week 54])
Description: Safety population that comprised of all participants who received at least one dose of study treatment were used for the assessment of serious adverse events and non-serious adverse events.
Arm/Group | Daprodustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/136 | 1/135
Serious Adverse Events (participants affected / at risk) | 21/136 | 37/135
Other Adverse Events (participants affected / at risk) | 102/136 | 102/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=136) | Darbepoetin Alfa (N=135)
Shunt stenosis (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=136) | Darbepoetin Alfa (N=135)
Nasopharyngitis (Infections and infestations) | 57 (110) | 73 (135)
Pharyngitis (Infections and infestations) | 10 (11) | 6 (6)
Gastroenteritis (Infections and infestations) | 7 (7) | 2 (2)
Shunt stenosis (Injury, poisoning and procedural complications) | 16 (30) | 15 (28)
Contusion (Injury, poisoning and procedural complications) | 17 (21) | 10 (12)
Skin abrasion (Injury, poisoning and procedural complications) | 10 (14) | 7 (7)
Procedural hypotension (Injury, poisoning and procedural complications) | 11 (16) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 20 (24) | 12 (15)
Vomiting (Gastrointestinal disorders) | 15 (20) | 11 (13)
Nausea (Gastrointestinal disorders) | 9 (10) | 11 (13)
Constipation (Gastrointestinal disorders) | 8 (10) | 6 (6)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (13)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (10)
Headache (Nervous system disorders) | 8 (8) | 6 (8)
Hypertension (Vascular disorders) | 5 (9) | 8 (8)
Pyrexia (General disorders) | 7 (8) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02969655/SAP_000.pdf
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02969655/Prot_001.pdf